CLINICAL TRIAL: NCT02201602
Title: Sulphonylurea Receptor Mutation and Responsiveness to Gliclazide - a Pilot Proof of Concept, Randomised Cross-over Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khoo Teck Puat Hospital (Other)
Responsible Party: Principal Investigator, Su Chi Lim, Senior Consultant, Khoo Teck Puat Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Gliclazide
Record Dates: First submitted 2014-07-22; First posted 2014-07-28 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes
Keywords: sulphonylureas; gliclazide; glibenclamide
MeSH Terms: conditions — Diabetes Mellitus | interventions — Gliclazide; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gliclazide (Experimental): Gliclazide, 80 mg tablet, half to maximal dose, 3 weeks
  Interventions: Drug: Gliclazide
- Glibenclamide (Active Comparator): Glibenclamide, 5 mg tablet, half to maximal dose, 3 weeks
  Interventions: Drug: Glibenclamide

INTERVENTIONS:
Drug: Gliclazide
  Other Names: Sun-Glizide; SIN09350P
  Arms: Gliclazide
Drug: Glibenclamide
  Other Names: Benil; SIN07284P
  Arms: Glibenclamide

SUMMARY:
Gliclazide has greater glucose lowering efficacy than glibenclamide among type 2 diabetes mellitus patients with minor haplotype (K23/A1369) at the KCNJ11/ABCC gene locations.

DETAILED DESCRIPTION:
Sulphonylurea (SU) is a glucose-lowering agent used widely to treat type 2 diabetes mellitus (T2DM). SU promotes insulin secretion from the pancreatic islet beta cell via binding and inhibition of the ATP-sensitive potassium (KATP) channel. The KATP channel is made up of two subcomponents, an inner Kir6.2 K+ channel (coded by the KCNJ11 gene) and an outer SU receptor 1 (SUR1) (coded by the ABCC8 gene). Although all SUs are mechanistically similar in terms of increasing insulin secretion, they bind to distinct regions of Kir 6.2 and SUR1 to exert their function. Different types of SU (e.g. tolbutamide, glibenclamide, glipizide, glimepiride and gliclazide) can therefore be grouped by their binding sites (A/B/A+B site) on the KATP channel [3]. Interestingly, the KCNJ11 E23K (rs5219) variant was shown to confer susceptibility to T2DM and the ABCC8 S1369A (rs757110) variant was found to be in complete linkage disequilibrium with it i.e. inherited together as a genetic block (haplotype). A recent in vitro molecular study suggested that the minor haplotype (K23/A1369) of KATP channel is sensitive to inhibition by gliclazide (binds to A-site) but not glibenclamide (binds to A+B site), and that the increased responsiveness to gliclazide was largely due to the A1369 allele. Understanding how the response to these two SUs may vary with the presence of the minor haplotype (K23/A1369) would therefore be beneficial for customization of patient treatment to achieve better clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age 21-65
* HbA1c >8.0% on two consecutive visits

Exclusion Criteria:

* Currently taking insulin at a regime more complex than basal insulin
* Not willing to perform self-blood glucose monitoring (SBGM)
* Renal impairment i.e. eGFR<50mls/min
* Pregnancy or unwilling to practice adequate contraception
* Taking other medications that may affect blood glucose e.g. systemic glucocorticoids.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Mean blood glucose level | 6 days

SECONDARY OUTCOMES:
Glycemic variability | 6 days
  Glycemic variability will be assessed using the EasyGV software (http://www.phc.ox.ac.uk/research/diabetes/software/easygv/) which is capable of calculating 10 different measures of glycemic variability from continuous glucose monitoring data, such as Standard Deviation (SD) and M-value, mean amplitude of glycemic excursions (MAGE).

CONTACTS AND LOCATIONS:
Overall Officials: Su Chi Lim, MBBS, PhD, Principal Investigator — Khoo Teck Puat Hospital
Locations (1):
- Khoo Teck Puat Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Gloyn AL, Weedon MN, Owen KR, Turner MJ, Knight BA, Hitman G, Walker M, Levy JC, Sampson M, Halford S, McCarthy MI, Hattersley AT, Frayling TM. Large-scale association studies of variants in genes encoding the pancreatic beta-cell KATP channel subunits Kir6.2 (KCNJ11) and SUR1 (ABCC8) confirm that the KCNJ11 E23K variant is associated with type 2 diabetes. Diabetes. 2003 Feb;52(2):568-72. doi: 10.2337/diabetes.52.2.568. PMID 12540637
- [Background] Hamming KS, Soliman D, Matemisz LC, Niazi O, Lang Y, Gloyn AL, Light PE. Coexpression of the type 2 diabetes susceptibility gene variants KCNJ11 E23K and ABCC8 S1369A alter the ATP and sulfonylurea sensitivities of the ATP-sensitive K(+) channel. Diabetes. 2009 Oct;58(10):2419-24. doi: 10.2337/db09-0143. Epub 2009 Jul 8. PMID 19587354